CLINICAL TRIAL: NCT03616496
Title: Assessment of 18F-Florbetaben Whole-body PET Imaging for the Comprehensive Detection of Cardiac and Extracardiac Sites of Amyloid Deposits
Brief Title: Assessment of 18F-Florbetaben Whole-body PET for the Detection of Cardiac and Extracardiac Sites of Amyloid Deposits
Acronym: CAPRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pierre Yves MARIE, Professor, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-004054-24
Record Dates: First submitted 2018-07-27; First posted 2018-08-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Amyloidosis
Keywords: PET imaging; Cardiac Amyloidosis; Florbetaben; Heart failure; Cardiology
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Heart Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ATTR amyloidosis patients (Experimental): Intervention by this arm: PET/CT with injection of Neuraceq [4 MegaBecquerel /Kilogram (MBq/kg)], blood and urine sampling for protein electrophoresis, bone scintigraphy
  Interventions: Drug: Neuraceq PET/CT imaging
- AL amyloidosis patients (Experimental): Intervention by this arm: PET with injection of Neuraceq (4 MBq/kg), blood and urine sampling for protein electrophoresis, bone scintigraphy
  Interventions: Drug: Neuraceq PET/CT imaging
- Control subjects with aortic stenosis (Active Comparator): Intervention by this arm: PET with injection of Neuraceq (4 MBq/kg), blood and urine sampling for protein electrophoresis, bone scintigraphy.
  Control subjects are patients with aortic stenosis and left ventricular hypertrophy treated by surgery or by Transcatheter Aortic Valve Implantation (TAVI)
  Interventions: Drug: Neuraceq PET/CT imaging

INTERVENTIONS:
Drug: Neuraceq PET/CT imaging — PET/CT with Neuraceq injection, blood and urine sampling for protein electrophoresis, bone scintigraphy for the three arm (if the exams are present in the patient's medical record and are less than 3 months old, they do not need to be repeated
  Other Names: Bone scintigraphy; Blood and urine sampling for protein electrophoresis

SUMMARY:
Although being classified as a rare disease, cardiac amyloidosis constitutes an increasing cause of heart failure, which is often overlooked and thus poorly managed. Amyloidosis involves deposits of light chain immunoglobulins in the immunoglobulin light chain amyloidosis (AL) type, but it may also be of a hereditary type in mutated transthyretin amyloidosis (ATTRm) or of a senile type in wildtype transthyretin forms (ATTRwt).

Myocardial biopsy remains a gold standard for definitive diagnosis but it is a traumatic technique which only provides information on a limited number of sampled sites.

Useful but not fully specific signs of cardiac amyloidosis may also be provided by Magnetic Resonance Imaging or MRI (delayed retention imaging) and echocardiography (longitudinal strain pattern).

Notwithstanding the above, relatively specific markers of amyloid plaques are now available in Positron Emission Tomography (PET). These markers are primarily fluorinated tracers which have been developed for the diagnosis of Alzheimer's disease. Two of these have already been the subject of feasibility studies in the setting of cardiac amyloidosis diagnosis, on a maximum of 10 amyloidosis patients but with very favorable results.

The hypothesis is that one of these two tracers, Florbetaben labelled with Fluorine-18-Florbetaben (18F-Florbetaben) used in the study, has sufficiently strong and prolonged binding kinetics at the level of the amyloid plaques to allow: (i) achieving whole-body PET recordings and thus, (ii) identifying not only cardiac amyloidosis but also extracardiac binding sites, particularly those readily accessible to biopsy sampling. This hypothesis has been strengthened by a recent case report illustrating the ability of whole-body florbetaben-PET to image not only cardiac but also extra-cardiac sites of amyloid deposits (Clin Nucl Med. 2017;42(1):50-3).

DETAILED DESCRIPTION:
In addition, distinctive imaging patterns pointing to amyloidosis may also be documented by other imaging techniques although insufficiently specific (e.g. decreased cardiac uptake of metaiodobenzylguanidine (MIBG), evocative pattern of delayed retention at Magnetic Resonance Imaging (MRI) or at strain echocardiography. Specific markers of amyloid plaques have been developed for the diagnosis of Alzheimer's disease and were initially labeled with carbon-11 and more recently, with fluor-18. Most of these markers have already been the subject of feasibility studies on limited numbers of amyloidosis patients (max 10) but with favorable results. In a previous pilot study, one of these tracers, the 18F-Florbetaben used in the present study-protocol, exhibited particularly slow kinetics, with differences in cardiac uptake between patients and controls still being documented as late as 80-min following injection. This uptake was also found to be somewhat lower in the 5 ATTR patients comparatively to the 5 AL patients. It may be hypothesized that 18F-Florbetaben has sufficiently slow and prolonged binding kinetics at the level of the amyloid plaques to allow: (i) achieving whole-body PET recordings with current recording times of 20 to 30 min and thus, (ii) identifying not only cardiac amyloidosis but also extracardiac binding sites, particularly those readily accessible to biopsy sampling. This hypothesis has just been strengthened by a recent case report, published by investigators involved in the present project and illustrating the ability of whole-body 18F-Florbetaben-PET to image not only cardiac but also various extracardiac sites of amyloid deposits.The proposed study would be the first in which the sample size would be sufficient to provide a credible assessment of the ability of PET, using an amyloid plaque tracer, to identify cardiac amyloidosis and with a possible separate analysis of ATTR and AL forms. Moreover, it would also constitute the first study involving an extensive use of whole-body PET imaging to assess the benefit of amyloidosis detection, not only at the cardiac level, but also at peripheral sites, especially those accessible for biopsy (tongue, rectum, salivary glands, carpal tunnel, liver, subcutaneous tissue, thyroid,...).

Being able to confirm or invalidate the diagnosis of cardiac amyloidosis in a non-invasive manner and by guiding biopsy sampling to the most active extracardiac sites would be a major step forward for these patients whose diagnosis is most often established too late, i.e. at an advanced stage of heart failure.

In the longer term,18F-Florbetaben whole-body PET could be helpful for the non-invasive monitoring of the evolution of cardiac as well as extracardiac sites of amyloid deposits under dedicated specific treatments (chemotherapies in AL forms and specific treatments currently under investigation for the AL forms). Such monitoring is still impossible today.

ELIGIBILITY:
Inclusion Criteria:

* For all study participants

  1. Person affiliated to or beneficiary of, a social security plan
  2. Person informed about study organization and having signed the informed consent
* For ATTR amyloidosis patients:

  1. left ventricular concentric hypertrophy with a diastolic septal thickness ≥ 15 mm at echography (as defined by the current distribution of this parameter in the ATTR patients involved in a French national cohort of the Henri Mondor Hospital),
  2. clearly positive bone scan (> mild cardiac uptake) and/or concordant results at pathology of cardiac or extra-cardiac sites (Congo red-positive deposits under crossed polarized light and immunohistochemical staining for transthyretin).
* For AL amyloidosis patients:

  1. left ventricular concentric hypertrophy with a diastolic septal thickness ≥ 13 mm at echography (as defined by the current distribution of this parameter in the AL patients involved in the French national cohort of the Henri Mondor Hospital),
  2. significant cardiac disease evidenced by an increase in plasma N-Terminal ProBNP (or BNP) and/or in troponin T (or I), corresponding to a Mayo clinic score ≥ 2 ,
  3. concordant results at pathology of cardiac or extra-cardiac sites (Congo red-positive deposits under crossed polarized light and immunohistochemical staining for κ and λ immunoglobulin light chains).
* For control subjects:

  1. History of surgical or Transcatheter Aortic Valve Implantation (TAVI)treatment of aortic stenosis
  2. Matching with amyloidosis patients according to gender and age (± 5 years).
  3. Cardiac hypertrophy with a diastolic septal thickness ≥ 15 mm at echography when matching with an ATTR patient and ≥ 13 mm when matching with an AL patient.

Exclusion Criteria:

1. Known allergy to the active substance and to any excipient for 18F-Florbetaben or for the bone scintigraphy radiotracer (99mTc-MDP)
2. Pregnancy, breastfeeding and woman of childbearing age without effective contraception
3. Person referred in articles L.1121-5 to L.1121-8 and L.1122-2 of the Public Health Code:

   * Pregnant, parturient or breastfeeding woman
   * Person deprived of liberty for judicial or administrative decision
   * Person under psychiatric care
   * Person admitted to health or social institution for other reasons than research
   * Minor person (non-emancipated)
   * Adult person under legal protection (any form of public guardianship)
   * Adult person incapable of giving consent and not under legal protection
4. No obvious cause of cardiac disease except for mild to moderate hypertension in all study subjects, for cardiac amyloidosis in the amyloidosis groups and for aortic stenosis in the control group
5. Impossibility of performing 18F-Florbetaben PET (agitated, confused patient, etc.).
6. Sever left ventricular dysfunction with an ejection fraction ≤ 35%
7. Severe hepatic or renal failure.
8. For control patients only: monoclonal gammopathy on a previous protein electrophoresis or ≥ mild cardiac uptake on a previous bone scintigraphy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Definitive diagnosis of cardiac ATTR- or AL-amyloidosis upon current diagnosis standard (including cardiac or extracardiac biopsies), | upon 24 months
  The diagnosis will be made with standard parameters (including cardiac or extracardiac biopsies), Importantly, a " control " population, including patients with left ventricular hypertrophy definitively unrelated to amyloidosis (even for low to mild forms) will be added for the analysis (this hypertrophy is mandatory for reaching a comparable partial volume effect than with amyloidosis patients when recording myocardial PET activity).

SECONDARY OUTCOMES:
To assess the diagnostic performance of whole-body PET/CT recordings, as reported in the main objective, to identify AL and ATTR amyloidosis individually. | upon 24 months
  Identical to the primary endpoint, except that the analyses will be planned separately for AL and ATTR amyloidosis.
To determine whether (18)F-florbetaben whole-body PET/CT images can reveal extracardiac areas with increased activity | upon 24 months
  Areas of abnormal (18)F-florbetaben uptake will be studied on whole-body PET/CT
To compare the cardiac kinetics of (18)F-florbetaben and an early myocardial retention index, within the first 10 minutes following injection, between patients with cardiac amyloidosis and the control population | upon 24 month
  Comparative analysis of the evolution of myocardial SUV (Standard Uptake Value) and TBRtarget-to-blood pool ratio) ( values and of an early myocardial retention index during the 10 minutes post-injection period in patients and controls
To determine whether most patients with true-positive MRI for cardiac amyloidosis | upon 24 month
  the comparison of the analysis will be made with myocardial tissue-to-background ratios (TBR) where the activities measured in SUV will be expressed relative to a mean blood background activity.
To assess the intra- and inter-observer agreements for the analysis of (18)F-florbetaben whole-body PET/CT images. | upon 24 month
  Intra-observer and inter-observer reproducibility measurements of SUV and TBR values obtained at cardiac and extracardiac sites from whole-body PET / CT images of 20 patients with amyloidosis (10 with Type AL and 10 with an ATTR type).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves MARIE, MD,PhD, Principal Investigator — CHRU de NANCY BRABOIS
Locations (1):
- Chru Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No